CLINICAL TRIAL: NCT04357262
Title: Resiliency in Total Joint Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Jeremy Gililland, Principle Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 129070
Record Dates: First submitted 2020-04-15; First posted 2020-04-22 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Osteoarthritis
Keywords: Total Hip Arthroplasty; Total Knee Arthroplasty; Patient Reported Outcomes; Resilience
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): No other non-standard of care activities will be performed
- Intervention (Experimental): Will be signed up for the automated text messaging program (StreaMD)
  Interventions: Other: StreaMD

INTERVENTIONS:
Other: StreaMD — Patients who are randomized to the intervention arm will be signed up for the automated text messaging program. Patients will receive automated text messages related to their surgery during the study period and can also ask questions through the text messages program, where automated messages will be sent based on the questions asked.
  Arms: Intervention

SUMMARY:
The investigators primary objective is to determine how does participation in StreaMD affect patient reported outcomes after Total Hip Arthroplasty (THA) or Total Knee Arthroplasty (TKA)?

DETAILED DESCRIPTION:
Osteoarthritis is a leading cause of disability in the US. By conservative estimates, about 54 million adults in the US have doctor-diagnosed arthritis. The number of people expected to have arthritis by the year 2040 is more than 78 million. Total joint arthroplasty is considered the treatment of choice for end-stage osteoarthritis. Currently, more than 1 million hip and knee replacements are performed each year in the US. By 2030, primary THR is projected to grow 171% and primary TKR is projected to grow by up to 189%, for a projected 635,000 and 1.28 million procedures, respectively. The incidence of pre-operative psychological distress in this group of patients is reported between 30% and 60% and preoperative psychological distress is associated with poorer pain and functional outcomes after surgery. Resilience, characterized by an ability to bounce back or recover from stress, is increasingly recognized as a psychometric property affecting many outcomes' domains including outcomes after TJA. Better resilience could improve patients overall satisfaction with the procedure.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 and older who are receiving a total hip or knee replacement.

Exclusion Criteria:

* Patients enrolled in the MyMobility study
* Patients who do not have cell phones with text messaging capability
* Non-English speaking patients

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2022-01-12 (Actual); Study Completion 2022-01-12 (Actual)

PRIMARY OUTCOMES:
Patient Reported Outcome Score (PROMIS) following THA or TKA | Follow Up Visits up to 2-Years
  Patient reported outcome will consist of the Patient-Reported Outcomes Measurement Information System (PROMIS)
Patient Reported Outcome Score (HOOS Jr.) following THA or TKA | Follow Up Visits up to 2-Years
  Patient reported outcome will consist of the hip disability and osteoarthritis outcome score (HOOS Jr.)
Patient Reported Outcome Score (KOOS Jr.) following THA or TKA | Follow Up Visits up to 2-Years
  Patient reported outcome will consist of the knee injury and osteoarthritis outcome score (KOOS Jr.)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Gililland, M.D., Principal Investigator — University of Utah
Locations (1):
- University of Utah Orthopaedic Center, Salt Lake City, Utah, United States